CLINICAL TRIAL: NCT03375099
Title: Comparison of Lethal Means Counseling and an Active Control Condition, With and Without Provision of Gun Locks for Improving Safe Storage of Personal Firearms Among National Guard Personnel
Brief Title: Comparison of Lethal Means Counseling and an Active Control Condition, With and Without Provision of Gun Locks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Mississippi (Other)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: CH2-17022105
Record Dates: First submitted 2017-11-13; First posted 2017-12-15 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Intentional Self-Harm by Other Specified Means
Keywords: Firearms; Guns; Suicide; Means Safety; Means Restriction; Lethal Means Counseling
MeSH Terms: conditions — Suicide | interventions — Health

STUDY DESIGN:
Intervention Model Description: 2 (Lethal Means Counseling vs Health and Stress Reduction) x 2 (Provision of free gun locks vs No gun locks)
Who Masked: Participant
Masking Description: Participants will not be informed of the nature of the conditions other than the one they are randomly assigned to receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lethal Means Counseling (Experimental): National Guard Personnel will receive a single 15-25 minute session of lethal means counseling. The session will focus on increasing the safety of current storage practices for personal firearms (e.g., storing unloaded in a secure location separate from ammunition) as well as planning to voluntarily and temporarily store firearms away from the home during any future hypothetical suicidal crisis. This intervention utilizes a motivational interviewing framework in an effort to remain sensitive to the views and culture of firearm owners.
  Interventions: Behavioral: Lethal Means Counseling
- Lethal Means Counseling plus Gun Locks (Active Comparator): National Guard Personnel will receive a single 15-25 minute session of lethal means counseling. The session will focus on increasing the safety of current storage practices for personal firearms (e.g., storing unloaded in a secure location separate from ammunition) as well as planning to voluntarily and temporarily store firearms away from the home during any future hypothetical suicidal crisis. This intervention utilizes a motivational interviewing framework in an effort to remain sensitive to the views and culture of firearm owners. Individuals in this condition will also receive a free gun (cable) lock for each of their personal firearms.
  Interventions: Behavioral: Lethal Means Counseling
- Health and Stress Reduction (Active Comparator): Individuals in this condition will take part in a single 15-25 minute session focused on reducing health vulnerabilities in one of four areas: diet, exercise, sleep, or stress. This condition is designed to control for the effects of active interaction with a clinicians (e.g. common factors). As with the experimental condition, this session will utilize a motivational interviewing framework.
  Interventions: Behavioral: Health and Stress Reduction
- Health + Stress Reduction plus Gun Locks (Active Comparator): Individuals in this condition will take part in a single 15-25 minute session focused on reducing health vulnerabilities in one of four areas: diet, exercise, sleep, or stress. This condition is designed to control for the effects of active interaction with a clinicians (e.g. common factors). As with the experimental condition, this session will utilize a motivational interviewing framework. Individuals randomized to this condition will also receive a free gun (cable) lock for each of their personal firearms. This will control for whether the effect of the provision of gun locks is accounted for by the simultaneous use of lethal means counseling.
  Interventions: Behavioral: Health and Stress Reduction

INTERVENTIONS:
Behavioral: Lethal Means Counseling — Single session motivational interviewing based interaction aimed to increase the safe storage of firearms in an effort to reduce suicide risk.
  Arms: Lethal Means Counseling; Lethal Means Counseling plus Gun Locks
Behavioral: Health and Stress Reduction — Single session motivational interviewing based interaction aimed to reduce vulnerability to negative outcomes across four domains: sleep, diet, exercise, and stress.
  Arms: Health + Stress Reduction plus Gun Locks; Health and Stress Reduction

SUMMARY:
In 2013, the National Guard reported a suicide rate that was substantially higher than both the general population and the active duty component of the United States military. The prototypical National Guard suicide decedent appears to be a young male firearm owner not currently deployed who dies using his own gun. Prior research within the military has revealed that soldiers are unlikely to seek out or engage in mental health services. In sum, current best practices in suicide risk assessment are poorly equipped to identify the individuals most likely to die by suicide. This study aims to examine the acceptability, feasibility, and utility of a single lethal means counseling session as part of a suicide prevention approach targeting demographic groups overrepresented in National Guard firearm suicides. 232 firearm-owning National Guard personnel will be randomized to one of four conditions, each of which requires a single 15-25 minute session: (1) lethal means counseling (2) lethal means counseling plus the provision of free gun locks (3) health and stress control condition (4) health and stress control condition plus the provision of free gun locks. The investigators anticipate that those who receive lethal means counseling will subsequently store their personal firearms more safely and report being more willing to store their firearms away from the home during any hypothetical future suicidal crisis. The overarching goal of each hypothesis is to examine the extent to which gun owning young male National Guard personnel at varying levels of suicide risk are willing to engage in means safety.

DETAILED DESCRIPTION:
In 2013, the National Guard reported a suicide rate that was substantially higher than both the general population and the active duty component of the United States military. The prototypical National Guard suicide decedent appears to be a young male firearm owner not currently deployed who dies using his own gun. Prior research within the military has revealed that soldiers are unlikely to seek out or engage in mental health services. In sum, current best practices in suicide risk assessment are poorly equipped to identify the individuals most likely to die by suicide. This study aims to examine the acceptability, feasibility, and utility of a single lethal means counseling session as part of a suicide prevention approach targeting demographic groups overrepresented in National Guard firearm suicides. The study will utilize a 2x2 Factorial Design: Intervention (Lethal Means Counseling, Health and Stress Control) X Gun-Lock (Provided, Not Provided). Participants will be 232 firearm owning National Guard personnel. Lethal Means Counseling comprises education on risk factors for suicide, information on preventative resources, and encouragement to store guns safely and to temporarily remove guns during high risk periods. The Health and Stress Program is designed to control for effects of general mental and physical health education in the active condition. Each condition utilizes a motivational interviewing framework. The overarching goal of each hypothesis is to examine the extent to which gun owning young male National Guard personnel at varying levels of suicide risk are willing to engage in safety planning and find means safety approaches acceptable

ELIGIBILITY:
Inclusion Criteria:

* Affiliated with the National Guard
* Owns at least one personal firearm
* Speaks English fluently

Exclusion Criteria:

* N/A

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 232 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Changes in Safe Storage of Personal Firearms | Change will be assessed at 3- and 6-month follow-up
  Whether firearms are stored (1) in a lock box or gun safe (yes/no) (2) loaded (yes/no) (3) separate from ammunition (yes/no) and (4) using a locking device (e.g. cable lock; yes/no)

SECONDARY OUTCOMES:
Perceived Cultural Competence and Likelihood of Effectiveness of Lethal Means Counseling [Acceptability and Perceived Utility] | This will be assessed immediately after the intervention at baseline
  Degree to which lethal means counseling is experienced as culturally respectful and likely to be beneficial
Changes in Willingness to Seek Mental Health Care in the Future | Change will be assessed immediately after the intervention and at 3- and 6-month follow-up
  Degree of openness to seeking future mental health care after receiving this intervention
Changes Openness to Means Safety in the Future | Change will be assessed immediately after the intervention and at 3- and 6-month follow-up
  Degree of openness to voluntarily and temporarily storing firearms away from the home during hypothetical future suicidal crises

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Anestis, PhD, Principal Investigator — Rutgers University
Locations (1):
- University of Southern Mississippi, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
We are open to collaborating with other researchers and making data available on an individual basis. No personally identifiable information would be included and we would first seek the approval of the funding agency (Military Suicide Research Consortium) due to their use of Common Data Elements.

REFERENCES:
- [Result] Anestis MD, Bryan CJ, Capron DW, Bryan AO. Lethal Means Counseling, Distribution of Cable Locks, and Safe Firearm Storage Practices Among the Mississippi National Guard: A Factorial Randomized Controlled Trial, 2018-2020. Am J Public Health. 2021 Feb;111(2):309-317. doi: 10.2105/AJPH.2020.306019. Epub 2020 Dec 22. PMID 33351652